CLINICAL TRIAL: NCT03674502
Title: A Phase 1 Study to Evaluate the Safety and Pharmacokinetics of ADU-1604, an Anti-CTLA-4 Antibody, in Adults With Metastatic Melanoma
Brief Title: Safety of ADU-1604 in Adults With Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to business realignment
Sponsor: Aduro Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADU-CL-17
Record Dates: First submitted 2018-09-11; First posted 2018-09-17 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ADU-1604 (Experimental): ADU-1604 administered as an IV infusion
  Interventions: Drug: ADU-1604

INTERVENTIONS:
Drug: ADU-1604 — anti-CTLA-4 monoclonal antibody

SUMMARY:
This study is a first-in-human, open-label, multicenter, dose-escalation study designed to evaluate the safety, PK, and PD of ADU-1604 and explore initial clinical activity in adults with metastatic melanoma.

DETAILED DESCRIPTION:
ADU-CL-17 is a first-in-human, open-label, multicenter, dose-escalation study designed to evaluate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of ADU-1604, an anti-CTLA-4 monoclonal antibody, and explore initial clinical activity in adults with metastatic melanoma. The primary objective of the study is to determine the Recommended Phase 2 Dose (RP2D) of ADU-1604 administered by IV infusion once every 3 weeks for 4 doses.

The study will be conducted in two parts: Dose Escalation followed by Dose Confirmation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years
2. Histologically-confirmed metastatic or unresectable melanoma
3. Progression of disease following at least one prior therapy, and is not a candidate for, or is intolerant to, established therapy known to provide clinical benefit (i.e. available treatment options have been exhausted). Subjects must have BRAF mutation status confirmed; if a subject is BRAF V600E/K positive, they must have received a BRAF- targeted regimen prior to entering the study, unless the patient was deemed ineligible for such treatment
4. Measurable disease according to RECIST (v1.1) [NOT required during Dose Escalation]
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Exclusion Criteria:

1. Prior diagnosis of uveal or mucosal melanoma
2. Prior treatment with CTLA-4-directed therapy in the metastatic setting. Use of CTLA- 4-directed treatment in the adjuvant or neoadjuvant setting is acceptable provided the last dose was >6 months before the first dose of ADU-1604 and there was no discontinuation of treatment due to a treatment-related toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Identify the recommended P2 dose (RP2D) of ADU-1604 administered as an IV infusion | 9 months

CONTACTS AND LOCATIONS:
Locations (5):
- France (3):
  - Hôpital de la Timone, Marseille
  - Hospital Saint Louis, Paris
  - Gustave- Roussy Institute, Villejuif
- Spain (2):
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No